CLINICAL TRIAL: NCT06526442
Title: Experimental and Clinical Study of Three-dimensional Magnetic Resonance Elastography to Evaluate Pancreatic Cancer and Interstitial Fibrosis
Brief Title: MRE for Diagnosis of Pancreatic Masses
Acronym: MREDPCM
Status: Recruiting | Type: Observational
Sponsor: Yu Shi (Other)
Responsible Party: Sponsor-Investigator, Yu Shi, Associate Professor, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Other Study IDs: SJ-16001-MRE
Record Dates: First submitted 2024-07-17; First posted 2024-07-29 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Neoplasm; Magnetic Resonance Imaging
Keywords: Pancreatic Cancer, solid pancreatic mass; Magnetic Resonance Elastography
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Plan to include patients with resectable pancreatic cancer 150: Investigators anticipate that 150 resectable pancreatic cancer participants are enrolled in this group and all participants undego magnetic resonance imaging.
  Interventions: Diagnostic Test: magnetic resonance imaging
- Plan to include patients with unresectable pancreatic cancer 50: Investigators anticipate that 50 unresectable pancreatic cancer participants are enrolled in this group and all participants undego magnetic resonance imaging.
  Interventions: Diagnostic Test: magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: magnetic resonance imaging — all participants undergo novel MR sequences, including 3D-MRE，DCE-MRI，IVIM-DWI，T1/T2 mapping.
  Other Names: MR elastrogaphy

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) accounts for 85-95% of pancreatic cancer and is one of the deadliest tumors in the world, with a survival rate of less than 8%, and identifying key prognostic or predictive factors facilitates risk stratification and prospective assessment in clinical trials. The extracellular matrix (ECM) surrounding PDAC often exhibits a large number of interstitial fibrosis, which is closely related to the formation, development and metastasis of PDAC. High order three-dimensional MR elastography (3D-MRE) allows non-invasive measurements of sheer stiffness in normal pancreas and pancreatic lesions. However, there are no reports about the application of MRE imaging biomarkers to predict the prognosis of PDAC at home and abroad.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) accounts for 85-95% of pancreatic cancer and is one of the deadliest tumors in the world, with a survival rate of less than 8%, and identifying key prognostic or predictive factors facilitates risk stratification and prospective assessment in clinical trials.

The extracellular matrix (ECM) surrounding PDAC often exhibits a large number of interstitial fibrosis, which is closely related to the formation, development and metastasis of PDAC. Although interstitial composition is considered a double-edged sword, influencing cancer biological progression and modification in multiple complex ways, experimental studies consistently demonstrate that hardening of ECM in PDAC accelerates PDAC progression and is significantly associated with shorter survival. If investigators can noninvasively detect the mechanical properties (hardness) of human PDAC before treatment, it will be helpful to describe the biological characteristics of tumors, predict the prognosis of patients, and choose the right clinical treatment decision.

High order three-dimensional MR elastography (3D-MRE) allows non-invasive measurements of sheer stiffness in normal pancreas and pancreatic lesions. However, there are no reports about the application of MRE imaging biomarkers to predict the prognosis of PDAC at home and abroad.

ELIGIBILITY:
Inclusion Criteria:

1. granting of written informed consent
2. age ≥18 years
3. no history of extrapancreatic malignancy
4. no preoperative biliary drainage
5. definitive histologic evidence of PDAC in excisional biopsy
6. with no less than three months of postoperative mortality or six months of follow- up

Exclusion Criteria:

1. inability to re-review of tissue specimens
2. unacceptable estimates of MRE parameters, specifically invalid wave data during postprocessing, inconsistent breath-holdings, intolerable pain, and MRE hardware disconnection
3. tumor diameters <1.0 cm
4. withdrawal/dropout during follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: participants aged 18-80 years
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Analyzing the measurement accuracy of MRE. | 9 months
  The hardness was measured by a hardness tester during the operation, and the mechanical parameters were measured by atomic force microscopy of the in vitro specimen. The measurement accuracy of MRE was analyzed by comparing the hardness tester and atomic force microscope results.
Radiological assessment of tumor stiffness. | 9 months
  A self-written script program in MATLAB is used to read and analyze mechanical group diagrams and waveform diagrams in three directions of x, y, and z, and a region of interest (ROI) delineation function is embedded.After drawing the ROI, an Excel file containing the corresponding values is automatically generated, and the average values of various mechanical parameters are calculated, including shear modulus (|G*|, SS), storage modulus (G', SM), loss modulus (G'', LM) and damping ratio (ӡ, DR).
Evaluation of tumor response to chemotherapy. | 12 months
  RECIST criteria (version 1.1) were used to objectively evaluate the response to chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Shi, MD.PhD., Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing hospital of china medical university, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang A, Gu C, Liu Y, Luo B, Zeng Y, Zhou M, Li C, Pan C, Wu L, Hu Z, Zhang X, Gao F, Shi Y. ITGB5-mediated biomechanical regulation in pancreatic ductal adenocarcinoma stroma impacts tumor progression and prognosis. J Transl Med. 2025 Oct 21;23(1):1150. doi: 10.1186/s12967-025-07119-5. PMID 41121153